CLINICAL TRIAL: NCT05976919
Title: Evaluating Treatable Traits Across the Spectrum of Chronic Obstructive Airways Disease
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Oliver Price, Principal Investigator, University of Leeds
Other Study IDs: 323694
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Airway Disease
MeSH Terms: interventions — Respiratory Function Tests; Exercise Test; Exercise; Absorptiometry, Photon; Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- COPD
  Interventions: Diagnostic Test: Pulmonary function testing
- Asthma
  Interventions: Diagnostic Test: Pulmonary function testing
- Bronchiectasis
  Interventions: Diagnostic Test: Pulmonary function testing
- Cystic fibrosis
  Interventions: Diagnostic Test: Pulmonary function testing
- Primary ciliary dyskinesia
  Interventions: Diagnostic Test: Pulmonary function testing

INTERVENTIONS:
Diagnostic Test: Pulmonary function testing — Physiological assessment of pulmonary physiology (large and small airways), exercise capacity, physical activity and body composition.
  Other Names: Cardiopulmonary exercise testing; Physical activity (daily step count); Dual-energy X-ray absorptiometry (body composition)

SUMMARY:
Respiratory disease affects one in five people and is a leading cause of global morbidity and mortality. Chronic obstructive airways diseases encompass conditions characterised by expiratory airflow limitation, exertional dyspnoea, activity limitation and impaired quality of life. The most common conditions include chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis, cystic fibrosis and primary ciliary dyskinesia. In recent years, there has been concerted effort in the scientific and respiratory medicine community to improve the diagnosis and management of chronic obstructive airways diseases using personalised or precision medicine (i.e., tailoring therapies and interventions according to specific "treatable traits") and identifying phenotypes or endotypes using validated biomarkers. To date, however, research in this setting has primarily focussed on people with COPD and asthma, with limited studies in other forms of chronic obstructive airways diseases. The aim of this study is therefore two-fold; first, to compare pulmonary physiology (i.e., large and small airway involvement) and extra-pulmonary manifestations across the spectrum of chronic obstructive airways, and second, to determine how disease-specific treatable traits associate with physical activity and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of airways disease in accordance with European Respiratory Society guidelines.
* Non / ex-smokers (packs recorded as cigarettes per day / years smoked).
* Male or female aged 18-65 years
* Ability to provide written informed consent.
* Full comprehension of spoken and written English language.
* Cystic Fibrosis patients on triple CFTR modulators (90% cohort)
* Cystic Fibrosis patients on no CFTR modulators
* Healthy controls - entirely asymptomatic, no prior history of inhaler medication use and free from respiratory disease.

Exclusion Criteria:

* Severe exacerbation requiring hospital admission or oral corticosteroids (OCS) in the past two months.
* Absolute or relative contraindications to cardio-pulmonary exercise testing or submaximal exercise testing.
* Absolute or relative contraindications to pulmonary function testing .
* Absolute or relative contraindications to dual energy x-ray (DEXA) scanning (i.e., pregnancy, recent contrast media administration or subject weight).
* Non-ambulant or musculoskeletal impairment that may affect activities of daily living or maximal exercise testing.
* Significant cognitive impairment (i.e., unable to provide written informed consent or safely / successfully perform tests).
* Currently receiving oxygen therapy.
* Inability to consent.
* Burkholderia Cepacia Complex, mycobacterium tuberculosis or mycobacterium abseccus infection.
* Lung transplantation
* Diagnosis of cardiovascular disease.
* Abnormal blood screening (anaemia, moderate / severe renal failure etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Chronic obstructive airways disease
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 7 day period
  Step-count

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No